## DOCUMENTO DE INFORMACIÓN PARA EL PARTICIPANTE

Título de la investigación:

Traducción y validación al español del BESTest y del mini BESTest

Nos dirigimos a usted para invitarle a participar en un proyecto de investigación que estamos realizando en la Universidad de Zaragoza y el Hospital Universitario Miguel Servet. Su participación es importante para obtener el conocimiento que necesitamos, pero antes de tomar una decisión debe:

- Leer este documento entero
- Entender la información que contiene el documento
- Hacer todas las preguntas que considere necesarias
- Tomar una decisión meditada
- Firmar el consentimiento informado, si finalmente desea participar.

Si decide participar se le entregará una copia de este documento y del consentimiento firmado. Por favor, consérvelos por si lo necesitara en un futuro.

Se le solicita su colaboración porque es usted una persona mayor de 65 años, sin problemas de salud destacables y autónomo para las actividades de la vida diaria. En total en el estudio participarán 12 personas con estas características.

Este estudio tiene por objetivo traducir y validar al español una escala de evaluación del equilibrio llamada BESTest y su versión abreviada, el mini BESTest, cuyo idioma original es el inglés.

Recuerde que su participación es voluntaria y consiste en llevar a cabo una evaluación pautada de su equilibrio durante algo más de una hora. Tendrá que realizar varias pruebas con las que valoraremos su equilibrio, todas ellas en una única sesión. Además del BEST y miniBESTest, completará las escalas de equilibrio de Berg, Escala de eficacia en caídas y el Test de levantarse y caminar. Se trata en todos los casos de valorar la calidad con la que usted es capaz de realizar transferencias, mantenerse de pie o desplazarse con diferentes niveles de dificultad. Los materiales necesarios para la evaluación (silla, rampa, cronómetro...) serán aportados por el examinador. La valoración se realizará de manera segura, evitando que usted pueda caerse.

Al tratarse de un estudio de investigación orientado a generar conocimiento usted no obtendrá ningún beneficio económico por su participación, si bien contribuirá al avance del conocimiento y al beneficio social.

Toda la información recogida se tratará conforme a lo establecido en la Ley Orgánica 15/99, de protección de datos de carácter personal. En la base de datos del estudio no se incluirán datos personales: ni su nombre, ni ningún dato que le pueda identificar. Se le identificará por un código que sólo el equipo investigador podrá relacionar con su nombre.

Para ejercer su derecho de acceso, rectificación, cancelación y oposición respecto a sus datos obtenidos durante el estudio debe ponerse en contacto con el investigador principal.

Las conclusiones del estudio se presentarán en congresos y publicaciones científicas pero se harán siempre con datos agrupados y nunca se divulgará nada que le pueda identificar.

Este proyecto no recibe financiación. El conocimiento derivado de este estudio puede generar en un futuro beneficios comerciales que pertenecerán al equipo investigador. Los participantes no tendrán derecho a reclamar parte de ese beneficio.

Usted tiene derecho a conocer los resultados del presente estudio, tanto los resultados generales como los derivados de sus datos específicos. También tiene derecho a no conocer dichos resultados si así lo desea. Por este motivo en el documento de consentimiento informado le preguntaremos qué opción prefiere. En caso de que desee conocer los resultados, el investigador le hará llegar los resultados.

Tal como se ha señalado, su participación es totalmente voluntaria, puede decidir no participar o retirarse del estudio en cualquier momento sin tener que dar explicaciones. Basta con que le manifieste su intención al investigador principal del estudio.

Si usted desea retirarse del estudio se eliminarán los datos recogidos hasta ese momento.

En caso de duda o para cualquier consulta relacionada con su participación puede ponerse en contacto con el investigador responsable, Da. Ma Pilar Domínguez Oliván,

| en el teléfono | 976765500 | extensión | 4964 | en | horario | de | mañanas | 0 | por | correo |
|---|---|---|---|---|---|---|---|---|---|---|
| electrónico en la | a dirección | mpdomi | n@uni | izar. | .es | | | | | |

Muchas gracias por su atención. Si finalmente desea participar le rogamos que firme el documento de consentimiento que se adjunta.

## **DOCUMENTO DE CONSENTIMIENTO INFORMADO**

| <b>Título del PROYECTO:</b> Traducción y validación al español del BESTest y del mini BESTest |
|---|
| Yo, (nombre y apellidos del participante) |
| He leído el documento de información que se me ha entregado. |
| He podido hacer preguntas sobre el estudio y he recibido suficiente información sobre el mismo. |
| He hablado con: Mª Pilar Domínguez Oliván |
| Comprendo que mi participación es voluntaria. |
| Comprendo que puedo retirarme del estudio: |
| 1) cuando quiera |
| 2) sin tener que dar explicaciones |
| 3) sin que esto repercuta en mis cuidados médicos |
| Presto libremente mi conformidad para participar en el estudio. |
| Deseo ser informado sobre los resultados del estudio: |
| sí no (marque lo que proceda) |
| He recibido una copia firmada de este Consentimiento Informado. |
| Firma del participante: |
| Fecha: |
| He explicado la naturaleza y el propósito del estudio al paciente mencionado Firma de la Investigadora: |
| Fecha: |